CLINICAL TRIAL: NCT04250987
Title: Exploratory Investigation of Data Obtained From a Sensor Connected to an Intermittent Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP304
Record Dates: First submitted 2020-01-21; First posted 2020-01-31 (Actual); Results first posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Compliance, Patient
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Intervention Model Description: Single arm - open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IC connected to a sensor (Experimental): Single use of a IC connected to a sensor
  Interventions: Device: SpeediCath(R)

INTERVENTIONS:
Device: SpeediCath(R) — IC SpeediCath ® connected to pressure sensor

SUMMARY:
The purpose of the investigational device in the proposed clinical investigation is to capture pressure data prior to and during voiding using a CE-marked commercially available catheter.

DETAILED DESCRIPTION:
This clinical investigation is based on an open explorative design evaluating the sensor ability to record readable data in healthy volunteers and the extent of artifacts influencing data quality and readability in healthy volunteers.

Overall:

* Single arm. Open-labelled, not randomized
* Healthy volunteers

Duration:

Information visit:

Oral and written information about the evaluation is given by the PI or his/her representative. Subjects can continue to visit 0, inclusion visit, the same day - if the subject has decided on participation and if practically possible.

Visit 0 - Inclusion visit:

Informed consent signed. Subjects can continue to visit 1 - test visit the same day - if practically possible.

Visit 1 - test visit:

1h test visit at Rigshospitalet. Fertile females will be asked to perform a pregnancy test. Subject is asked about symptoms for urinary tract infections (frequent urination, stinging or pain at urination). If negative for these symptoms, the subject will be catheterised with (SpeediCath® Standard, male/female, Nelaton tip depending of the gender) with fitted pressure sensor. The urine is led into a standard urine flowmeter.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Be at least 18 years of age and have full legal capacity

Exclusion Criteria:

1. Previous history of genitourinary disease in-cluding congenital abnormalities and surgical procedures performed in the urinary tract
2. Symptoms of urinary tract infections (fre-quent urination, stinging and pain at urina-tion)
3. Participation in any other clinical investiga-tions during this investigation (Inclusion → termination)
4. Known hypersensitivity toward any of the test products
5. Positive pregnancy tes for women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — at least 4 of each gender
Enrollment: 12 (Actual)
Dates: Start 2019-03-23 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Ceder, M.Sc, Study Director — Head of Clinical Operations
Locations (1):
- Department of Urology, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Undergoing Catheterization With SpeediCath ®: One time use of intermittent catheterization with SpeediCath ® connected to a pressure sensor for 8 males and 4 females
Period: Overall Study
Arm/Group | Participants Undergoing Catheterization With SpeediCath ®
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: One time use of intermittent catheterization with SpeediCath ® connected to a pressure sensor for 8 males and 4 females
Arm/Group | Participants Undergoing Catheterization With SpeediCath ®
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Denmark | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Readability of Pressure Sensor Measurements
Description: Determination of whether the sensor could detect changes in pressure in kilopascal (kPa) and provide a readable graph depicting changes in kPa over time of use of IC. Each pressure sensor graph is assessed visually to determine whether the instrument can be used in future studies on a Yes/No basis. The total number of participants with readable pressure sensor measurements were counted.
Time Frame: 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Undergoing Catheterization With SpeediCath ®
Number analyzed (Participants) | 12
Participants | 11

ADVERSE EVENTS:
Time Frame: 1 hour
Arm/Group | Participants Undergoing Catheterization With SpeediCath ®
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-30): https://cdn.clinicaltrials.gov/large-docs/87/NCT04250987/Prot_SAP_000.pdf